CLINICAL TRIAL: NCT00462566
Title: The Efficacy of Motor Cortex Stimulation for Pain Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Dalhousie University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CDHA004
Record Dates: First submitted 2007-04-17; First posted 2007-04-19 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-06

CONDITIONS: Neuropathic Pain; Phantom Limb Pain; Stump Pain; Brachial Plexus Avulsion; Deafferentation Pain; Facial Pain; Complex Regional Pain Syndrome
Keywords: Motor cortex stimulation; neuropathic; pain; complex regional pain syndrome; deafferentation facial pain
MeSH Terms: conditions — Neuralgia; Phantom Limb; Causalgia; Facial Pain; Complex Regional Pain Syndromes; Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: motor cortex stimulation

SUMMARY:
The objective is to determine if motor cortex stimulation works for the following conditions:

1. Deafferentation facial pain,
2. Upper extremity complex regional pain syndrome (CRPS) and
3. Brachial plexus avulsion or phantom limb pain.

Each of these groups of 6 patients (total of 18) will be studied independently and all patients will be implanted with a motor cortex stimulation system. They will be randomised to either a regular or low stimulation setting in the two arms of the study. Each arm will last 3 months.

DETAILED DESCRIPTION:
This is a prospective, blinded randomized crossover study comparing two stimulation paradigms in three different groups of patients receiving motor cortex stimulation. The aim of this study is to examine the effectiveness of this modality in a controlled blinded manner, which has not been done in previous studies. There are two primary purposes of this study. The first is to compare two different stimulation paradigms: "high" level stimulation (i.e. stimulator activated 'on' for 10 minutes, 'off' for 2 hours; presumed therapeutic dose); versus "low" stimulation ('on' for 1 minute, 'off' for 6 hours; presumed subtherapeutic dose), in a prospective blinded crossover study design.

The second purpose of this study, is to examine the outcome of MCS in three different pain groups. These are:

1. Unilateral upper extremity neuropathic pain such as brachial plexus avulsion, stump pain or phantom limb pain
2. Neuropathic deafferentation facial pain
3. Upper extremity complex regional pain syndrome (CRPS)

Measurements of the effects of motor cortex stimulation will include a visual analogue scale (VAS) of perceived pain, the McGill Pain Questionnaire, SF-36 quality of life questionnaire, Beck Depression Inventory-II, the standard 7-point patient global impression of change (PGIC), medications log (verified by pharmacy records) and an employment status questionnaire. Adverse events will be recorded at each visit.

Table 1:

Visit Study Week Standard Care 0a 1b 12c 24d 1a 2e 3f 4g F/Uh Clinic Visit X X X X X X Consent X Surgery X X X Program MCS X X X X X X VAS X X X X X X X SF-36 X X X X X X X Medications Log X X X X Employment Status X X X X McGill Pain X X X X X X X Beck Depression II X X X X Global impression of change X X

1. Screening visit in consideration of MCS
2. Immediate post-op visit, randomization to high or low settings
3. 12 week crossover point
4. Final study visit, MCS programmed at 'best' settings
5. Trial period of MCS, lasting for 1 to 2 weeks
6. Clinic visit to determine efficacy of MCS and removal of temporary external system.
7. Permanent implantation of MCS, if trial was successful
8. Follow-up as required.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis in one of the following three categories:

   * Unilateral upper extremity neuropathic pain such as phantom limb pain, stump pain or brachial plexus avulsion
   * Neuropathic deafferentation facial pain
   * Upper extremity complex regional pain syndrome (CRPS)
2. Pain is refractory to conservative methods (e.g. medications, regional blocks) as reviewed by a chronic pain clinical physician
3. Patient is considered a good candidate for neurosurgery, i.e. no other medical problems that would preclude surgery
4. Patients who are willing to provide informed consent.

Exclusion Criteria:

1. Patients who are not considered medically fit for neurosurgery.
2. Patients who have not exhausted conservative methods of pain control, prior to considering motor cortex stimulation.
3. Patients who are not able to provide informed consent.
4. Patients unable to have magnetic resonance imaging (MRI).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Visual Analog scale | 1 month preop, at 12 and 24 weeks postop
SF-36 | 1 month preop, at 12 and 24 weeks postop
McGill Pain questionnaire | 1 month preop, at 12 and 24 weeks postop
Beck II depression | 1 month preop, at 12 and 24 weeks postop
Global impression of change | at 12 and 24 weeks postop
Medications log | 1 month preop, at 12 and 24 weeks postop
Employment status | 1 month preop, at 12 and 24 weeks postop

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Brownstone, MD, PhD, Principal Investigator — Dalhousie University, Queen Elizabeth II Health Sciences Centre
Locations (1):
- Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia, Canada

REFERENCES:
- [Result] Radic JA, Beauprie I, Chiasson P, Kiss ZH, Brownstone RM. Motor Cortex Stimulation for Neuropathic Pain: A Randomized Cross-over Trial. Can J Neurol Sci. 2015 Nov;42(6):401-9. doi: 10.1017/cjn.2015.292. Epub 2015 Sep 1. PMID 26324857